CLINICAL TRIAL: NCT00971724
Title: A Randomized, Placebo-controlled, Double-blind, Single-center Study Using Multiple Doses of Prednisolone to Quantify Effects on Selected Biomarkers and Assess Pharmacokinetics in Healthy Males
Brief Title: Biomarkers of Prednisolone Treatment (P05888)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P05888; 294001 (Other: Merck)
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Insulin Resistance; Hyperglycemia; Glucose Intolerance
Keywords: Prednisolone; Glucocorticoids
MeSH Terms: conditions — Insulin Resistance; Hyperglycemia; Glucose Intolerance | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo (Placebo Comparator): Treatment with placebo for 15 days
  Interventions: Drug: Placebo
- Prednisolone 7.5 mg daily (Experimental): Treatment with prednisolone 7.5 mg daily for 15 days
  Interventions: Drug: Prednisolone
- Prednisolone 15 mg daily (Experimental): Treatment with prednisolone 15 mg daily for 15 days
  Interventions: Drug: Prednisolone
- Prednisolone 30 mg daily (Experimental): Treatment with prednisolone 30 mg daily for 15 days
  Interventions: Drug: Prednisolone
- Prednisolone 75 mg (Experimental): Treatment with prednisolone 75 mg for a single day
  Interventions: Drug: Prednisolone
- Prednisolone 15 mg twice daily (Experimental): Treatment with prednisolone 15 mg twice daily for a single day
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Placebo — Oral administration, once daily, for 15 days
  Arms: Placebo
Drug: Prednisolone — Oral administration
  Arms: Prednisolone 15 mg daily; Prednisolone 15 mg twice daily; Prednisolone 30 mg daily; Prednisolone 7.5 mg daily; Prednisolone 75 mg

SUMMARY:
Primary objective:

* To identify a biomarker or biomarker-set for the adverse metabolic effects of various doses of prednisolone treatment.

Secondary objectives:

* To describe the PK of prednisolone and PD of a series of biomarkers.
* To identify biomarkers that reflect side effects of prednisolone.
* To elucidate part of the mechanisms by which prednisolone induces metabolic changes.

ELIGIBILITY:
Inclusion Criteria:

* 22 < BMI < 30
* fasting glucose < 5.6 mmol/L and glucose < 7.8 mmol/L 2hr after OGTT
* able and willing to sign informed consent
* history of good physical and mental health
* subject smokes less than 5 cigarettes per day
* able to keep a normal day and night rhythm

Exclusion Criteria:

* allergy to prednisolone
* glucocorticoid use during last 3 months prior to study
* use of any drug or substance
* history of familiar diabetes type 2
* clinically relevant history or presence of any medical disorder
* clinically relevant abnormal lab or ECG
* positive drug or alcohol screen, positive hepatitis B or C surface antigen
* donation of blood (>100 mL) within 90 days prior to the first dose

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2006-05; Primary Completion 2006-10 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
To identify a biomarker or biomarker-set for adverse metabolic effects of various doses of prednisolone | Day 1 and day 15

SECONDARY OUTCOMES:
To describe the PK of prednisolone and PD of a series of biomarkers | Day 1 and day 15

REFERENCES:
- [Derived] Ellero-Simatos S, Szymanska E, Rullmann T, Dokter WH, Ramaker R, Berger R, van Iersel TM, Smilde AK, Hankemeier T, Alkema W. Assessing the metabolic effects of prednisolone in healthy volunteers using urine metabolic profiling. Genome Med. 2012 Nov 30;4(11):94. doi: 10.1186/gm395. eCollection 2012. PMID 23199229
- [Derived] Toonen EJ, Fleuren WW, Nassander U, van Lierop MJ, Bauerschmidt S, Dokter WH, Alkema W. Prednisolone-induced changes in gene-expression profiles in healthy volunteers. Pharmacogenomics. 2011 Jul;12(7):985-98. doi: 10.2217/pgs.11.34. Epub 2011 Jun 2. PMID 21635145